CLINICAL TRIAL: NCT06302738
Title: PhenotypIsatioN of Sleep Pattern in hyperTensive Patients With blOod Pressure Non-DIPper Status
Brief Title: Phenotypisation of Sleep Pattern in Hypertensive Patients With Non Dipper Pattern
Acronym: INTO-DIP
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C221
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Hypertension; Sleep Disorder
MeSH Terms: conditions — Hypertension; Sleep Wake Disorders | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-dipper pattern at 24-hour BP monitoring: Defined as a nocturnal decrease systolic and/or in diastolic BP values <10% compared to the corresponding daytime values;
  Interventions: Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: polysomnography — patients will undergo a home sleep study to evaluate the presence of sleep disorders

SUMMARY:
High blood pressure is the most common modifiable risk factor for cardiovascular diseases (CV). The large interindividual variability in clinical expression of the disease and response to treatment, however, makes the management of the hypertensive patient complex.Therefore, identifying phenotypes of hypertensive patients associated with a specific CV outcome or who tend to respond/not respond to treatment is of paramount importance for improving CV prevention.

It has been shown that the phenotype of hypertensive patient with poor control of nighttime blood pressure values, especially when associated with a "non-dipper" profile, was associated with an increased risk of developing CV and cerebrovascular complications.

The non-dipper profile and nocturnal hypertension are caused by several factors including excessive salt intake and dysautonomia. However, they are also inevitably influenced by sleep duration and the presence of sleep disorders: obstructive sleep apnea (OSA), but also insomnia and periodic movements of the lower limbs,such as those frequently seen in restless legs syndrome, are among the the main determinants related to altered nighttime pressure pattern. However, such disturbances are not systematically assessed during the performance of monitoring 24h pressor and their impact in the outcome of the hypertensive patient is unknown.

The primary objective of this study is to phenotype non-dipper patients with or without nocturnal hypertension to determine the prevalence of sleep disorders such as sleep apnea syndrome, insomnia, and restless legs syndrome (RLS) (OSA diagnosed considering AHI>5 events/hour, insomnia and RLS according to ICSD 3 criteria) and correlate the presence of various sleep disorders with cardiac organ damage, vascular, and renal damage mediated by hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old;
* arterial hypertension defined as: a) office systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg AND either 24-hour ambulatory systolic BP ≥130 mmHg and/or diastolic BP ≥80 mmHg OR b) the presence of antihypertensive treatment;
* non-dipper pattern at 24-hour BP monitoring (confirmed on repeated ABPM including one performed within 3 months prior to enrolment and one after enrolment, both on the same antihypertensive treatment, if any), defined as a nocturnal decrease systolic and/or in diastolic BP values <10% compared to the corresponding daytime values;
* signed written informed consent;

Exclusion Criteria:

* shift workers
* atrial fibrillation/flutter;
* pregnancy and lactation;
* terminal malignant disease, life expectancy <6 months;
* limb amputation;
* dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-dipper status with or without nocturnal hypertension
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disorders | baseline
  Phenotype patients with non-dipper status with or without nocturnal hypertension in order to establish the prevalence of sleep disturbances such as sleep apnea syndrome, insomnia and restless legs syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (11):
- Italy (11):
  - UOSD Ipertensione Arteriosa "A.M. Pirrelli" - AUOC Policlinico di Bari, University of Bari,, Bari, Italy, Bari
  - Azienda Sanitaria Locale della provincia di Brindisi, Brindisi, Italy, Brindisi
  - Medicina Interna 1, Ambulatorio Ipertensione e Malattie Metaboliche AOU "Maggiore della carità"- Novara, Novara, Italy, Novara
  - Padova 1- Clinica Medica 3 · Dipartimento di Medicina · Azienda Ospedaliera di Padova, Italy, Padua, Italy, Padova
  - Padova 2 - UOC Medicina d'urgenza, Centro Regionale Specializzato per l'ipertensione arteriosa OSA - Azienda ospedaliera Università di Padova, Italy, Padua, Italy, Padova
  - UO Cardiologia, UO Pneumologia, Presidio Ospedaliero Cittadella, Azienda ULSS 6 Euganea, Cittadella, Italy., Cittadella, Italy, PD
  - Azienda Unità Sanitaria Locale-IRCCS di Reggio Emilia- S.O.S Centro per la Cura dell'Ipertensione Arteriosa- Medicina II Cardiovascolare, Reggio Emilia, Italy, RE
  - Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento- UO Medicina interna - Rovereto, Rovereto, Italy, Trento
  - Azienda sanitaria universitaria Giuliano-Isontina (ASU-GI)- SC (UCO) Medicina Clinica, Trieste, Italy, Trieste
  - Department of Medicine, University of Verona, Verona, Italy, Verona, Italy, Verona
  - Istituto Auxologico Italiano IRCCS, Milan, MI